CLINICAL TRIAL: NCT03431532
Title: Neuraxial Versus General Anesthesia for Total Knee Replacement Surgery - Are There Different Effects on the Immune System?
Brief Title: Monocyte Subsets Altered by Anesthesia
Status: Completed | Type: Observational
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Other Study IDs: NA vs GA Immunology
Record Dates: First submitted 2018-01-30; First posted 2018-02-13 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2018-02

CONDITIONS: Regional Anesthesia; General Anesthesia; Immune Function
Keywords: anesthesia; general anesthesia; neuraxial anesthesia; monocyte funtion; CD 14, HLA-DR; Interleukines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neuraxial anesthesia: Patients with total knee replacement surgery having neuraxial anesthesia along with the procedure.
- general anesthesia: Patients with total knee replacement surgery having General anesthesia along with the procedure.

SUMMARY:
The impact of different anesthetic techniques on the immune system remains unclear.

Aim of this ex vivo / in vitro study was to determine the effects of general and neuraxial anesthesia on monocyte subset alteration and the release of prototypical pro- and anti-inflammatory cytokines. Twenty patients undergoing total knee replacement surgery were randomly assigned to receive either general anesthesia (ITN) or combined spinal/epidural anesthesia (CSE). CD14 and HLA-DR expression patterns on monocytes and intracellular TNF-alpha production were quantified via flow cytometry. TNF-α and IL-10 release were measured via enzyme linked immunosorbent assay (ELISA).

DETAILED DESCRIPTION:
Numerous of factors affect the immunological response during surgery. Despite intensive research, the impact of different anesthetic techniques on the immune system remains unclear.

Aim of this ex vivo / in vitro study was to determine the effects of general and neuraxial anesthesia on monocyte subset alteration and the release of prototypical pro- and anti-inflammatory cytokines. Twenty patients undergoing total knee replacement surgery were randomly assigned to receive either general anesthesia (ITN) or combined spinal/epidural anesthesia (CSE). Samples of venous blood were taken from the patients before and after induction of anesthesia, immediately, 6 hours, 24 hours, and 48 hours after surgery. All blood samples were incubated in presence or absence of LPS (lipopolysaccharide; 1 µg/ml) for 24 hours. CD14 and HLA-DR expression patterns on monocytes and intracellular TNF-alpha production were quantified via flow cytometry. TNF-α and IL-10 release were measured via enzyme linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Total knee replacement surgery
* 18 years or older

Exclusion Criteria:

* clinical signs of infection,
* neoplasia
* treatment with immunomodulatory agents
* any kind of immune mediated disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients ungergoing total knee replacement surgery in neuraxial or General aneshtesia
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
CD 14 and HLA-DR Expression Patterns on monocytes | 1 year
  CD 14 and HLA-DR Expression Patterns on monocytes in whole blood culture assay

SECONDARY OUTCOMES:
Intracellular TNF-alpha production | 1 year
  Intracellular TNF-alpha production in whole blood culture assay
TNF-alpha and IL-10 release | 1 year
  TNF-alpha and IL-10 release in whole blood culture assay

CONTACTS AND LOCATIONS:
Overall Officials: Sven Schneider, MD, Principal Investigator — Universität des Saarlandes
Locations (1):
- Sven O. Schneider, MD, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bomberg H, Volk T, Biedler A, Schneider SO. Impact of intraoperative blood salvage on monocyte subsets alteration and intracellular tumor necrosis factor-alpha production. J Biomed Mater Res A. 2018 Mar;106(3):815-821. doi: 10.1002/jbm.a.36281. Epub 2017 Nov 28. PMID 29094483
- [Background] Schneider SO, Rensing H, Hartmann L, Grundmann U, Volk T, Biedler A. Impact of intraoperatively salvaged and washed blood on stimulated cytokine release in vitro. Transfusion. 2014 Oct;54(10 Pt 2):2782-90. doi: 10.1111/trf.12781. Epub 2014 Oct 7. PMID 25294235
- [Background] Schneider SO, Biedler AE, Behmenburg F, Volk T, Rensing H. Impact of shed blood products on stimulated cytokine release in an in vitro model of transfusion. Acta Anaesthesiol Scand. 2012 Jul;56(6):724-9. doi: 10.1111/j.1399-6576.2012.02704.x. Epub 2012 May 9. PMID 22571497
- [Background] Schneider SO, Rensing H, Graber S, Kreuer S, Kleinschmidt S, Kreimeier S, Muller P, Mathes AM, Biedler AE. Impact of platelets and fresh frozen plasma in contrast to red cell concentrate on unstimulated and stimulated cytokine release in an in vitro model of transfusion. Scand J Immunol. 2009 Aug;70(2):101-5. doi: 10.1111/j.1365-3083.2009.02278.x. PMID 19630915
- [Background] Biedler AE, Schneider SO, Seyfert U, Rensing H, Grenner S, Girndt M, Bauer I, Bauer M. Impact of alloantigens and storage-associated factors on stimulated cytokine response in an in vitro model of blood transfusion. Anesthesiology. 2002 Nov;97(5):1102-9. doi: 10.1097/00000542-200211000-00011. PMID 12411792